CLINICAL TRIAL: NCT02682030
Title: Utilization of Pulmonary Clearance Devices in Amyotrophic Lateral Sclerosis
Brief Title: The Use of Airway Clearance Devices in ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Ashraf Elsayegh, Assistant Clinical Professor, UCLA School of Medicine, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00039699
Record Dates: First submitted 2016-02-04; First posted 2016-02-15 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Airway Clearance Devices; High Frequency Chest Compression Devices; Cough Assist
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment group A (Active Comparator): Subjects randomized to group A will be fitted for and issued a mechanical High Frequency Chest Compression Device (HFCC) device for home use. Subjects will be instructed to use the HFCC device 2-3 times per day for 15-30 minutes each. Subjects will be instructed to keep a device usage, concomitant medication, and adverse event diary.
  Interventions: Device: High Frequency Chest Compression Device (HFCC)
- Treatment group B- HFCC and Cough Assist (Active Comparator): Subjects randomized to group B will be fitted for and issued a mechanical High Frequency Chest Compression Device (HFCC) device and will also be issued a cough assist device. Subjects will be instructed in the use of both devices. The HFCC device should be utilized 2-3 times per day for 15-30 minutes each followed by a session with the cough assist. Subjects will be instructed to keep a device usage, concomitant medication, and adverse event diary.
  Interventions: Device: High Frequency Chest Compression Device (HFCC); Device: Cough Assist

INTERVENTIONS:
Device: High Frequency Chest Compression Device (HFCC) — A vest designed to help clear the airway of mucus and other secretions through mechanical knocking of the chest area.
Device: Cough Assist — A device that aids patients to clear mucus and secretions that they would otherwise be unable to clear with coughing.
  Arms: Treatment group B- HFCC and Cough Assist

SUMMARY:
The investigator is examining the use of one airway clearance medical device compared to the use of two airway clearance medical devices together in patients with amyotrophic lateral sclerosis (ALS). More specifically, the investigator wants to know how effective the use of either a mechanical High Frequency Chest Compression (HFCC) device is on its own or the use of both a mechanical High Frequency Chest Compression (HFCC) device and Cough Assist together to maintain a healthy airway and clear secretions.

The first device is a passive form of mechanical High Frequency Chest Compression (HFCC), which was designed to help clear the airway of mucus and other secretions through mechanical knocking of the chest area. The second device, called a Cough Assist, aids patients to clear mucus and secretions that they would otherwise be unable to clear with coughing. This study will enroll up to 20 people in total at CSMC.

DETAILED DESCRIPTION:
This 180 day (25.7 weeks) pilot study is designed to evaluate the effectiveness of airway clearance devices in adults with ALS. Subjects will be randomized in a 1:1 ratio to one of two treatment groups: treatment with a mechanical HCFF device alone or treatment with both a mechanical HFCC device and a cough assist device.

This outpatient study includes a screening/baseline visit followed by a 180 day (25.7 weeks) treatment period with three scheduled clinic visits (day 30, day 90, day 180). Pulmonary assessments and ALS outcome measures will be collected at each visit in addition to quality of life assessments and device usage diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected, possible, probable, Probable (Lab-Supported), or Definite ALS according to El Escorial Criteria
2. Males and females age 18 and above
3. Novel to airway clearance device use
4. Forced vital capacity ≤ 75% of predicted

Exclusion Criteria:

1. Any contraindication for pulmonary ventilation scan including allergy to radioisotopes
2. Any contraindication for use of a pulmonary clearance device

   * Susceptibility to pneumothorax
   * Recent (within 30 days) barotrauma
   * Unstable head or neck injury
   * Active hemorrhage with hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Elsayegh, MD, FCCP, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited internally at Cedars-Sinai Medical Center ALS multidisciplinary clinic.
Pre-assignment Details: 5 participants met inclusion criteria and were enrolled into the study. One participant was randomized to the Treatment Group A HFCC Only arm while 4 participants were randomized to the Treatment Group B HFCC + Cough Assist Arm.
Groups:
- Treatment Group A - HFCC Only: Subjects randomized to group A will be fitted for and issued a mechanical High Frequency Chest Compression Device (HFCC) device for home use. Subjects will be instructed to use the HFCC device 2-3 times per day for 15-30 minutes each. Subjects will be instructed to keep a device usage, concomitant medication, and adverse event diary.
  High Frequency Chest Compression Device (HFCC): A vest designed to help clear the airway of mucus and other secretions through mechanical knocking of the chest area.
Period: Overall Study
Arm/Group | Treatment Group A - HFCC Only | Treatment Group B- HFCC and Cough Assist
Started | 1 | 4
Completed | 0 | 2
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Subjects randomized to group A will be issued a mechanical High Frequency Chest Compression Device (HFCC) device for home use. Subjects randomized to group B will be issued a mechanical High Frequency Chest Compression Device (HFCC) device and will also be issued a cough assist device. Please see Baseline Characteristics for more information.
Groups:
- Treatment Group A HFCC Only: Subjects randomized to group A will be fitted for and issued a mechanical High Frequency Chest Compression Device (HFCC) device for home use. Subjects will be instructed to use the HFCC device 2-3 times per day for 15-30 minutes each. Subjects will be instructed to keep a device usage, concomitant medication, and adverse event diary.
  High Frequency Chest Compression Device (HFCC): A vest designed to help clear the airway of mucus and other secretions through mechanical knocking of the chest area.
- Treatment Group B HFCC + Cough Assist: Subjects randomized to group B will be fitted for and issued a mechanical High Frequency Chest Compression Device (HFCC) device and will also be issued a cough assist device. Subjects will be instructed in the use of both devices. The HFCC device should be utilized 2-3 times per day for 15-30 minutes each followed by a session with the cough assist. Subjects will be instructed to keep a device usage, concomitant medication, and adverse event diary.
  High Frequency Chest Compression Device (HFCC): A vest designed to help clear the airway of mucus and other secretions through mechanical knocking of the chest area.
  Cough Assist: A device that aids patients to clear mucus and secretions that they would otherwise be unable to clear with coughing.
- Total: Total of all reporting groups
Arm/Group | Treatment Group A HFCC Only | Treatment Group B HFCC + Cough Assist | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Continuous [Mean (Full Range); unit: years] | 78 [78 to 78] | 61.5 [49 to 81] | 64.8 [49 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 5
Height [Mean (Full Range); unit: centimeters] | 183 [183 to 183] | 173.25 [157 to 188] | 178.125 [157 to 188]
Weight [Mean (Full Range); unit: kilograms] | 87 [87 to 87] | 81.15 [68 to 88] | 84.075 [68 to 88]
Forced Vital Capacity [Mean (Full Range); unit: % Predicted] | 43 [43 to 43] | 64.25 [19 to 111] | 53.625 [19 to 111]
Forced Expiratory Volume [Mean (Full Range); unit: % Predicted] | 53 [53 to 53] | 67.5 [22 to 114] | 60.25 [22 to 114]
Maximum Inspiratory Pressure (MIP) [Mean (Full Range); unit: cm/H20] | 59 [59 to 59] | 72.25 [49 to 95] | 65.625 [45 to 95]
Maximum Expiratory Pressure (MEP) [Mean (Full Range); unit: cm/H20] | 27 [27 to 27] | 60 [17 to 104] | 43.5 [17 to 104]
Diffusion Capacity [Mean (Full Range); unit: ml/mmHg/min] | 12.7 [12.7 to 12.7] | 18.9 [14.8 to 23.1] | 15.8 [12.7 to 23.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Improved Respiratory Symptoms as Shown by Chest X-Ray Between Baseline and End of Study
Description: A projection radiograph of the chest used to diagnose conditions affecting the chest. Chest X-Ray performed at each study visit. Investigator looked at clinical impression of Chest X-ray to be normal versus abnormal. If there was presence of atelectasis, this indicated a worsening of subject's respiratory symptoms. If subject's Chest X-Ray impression remained the same and continually normal, this indicated no change in respiratory symptoms.
Time Frame: 1 time at screening/baseline and then at the month 1, month 3, and month 6 study visit for a total of 4 X-rays over 6 months.
Population: Chest X-ray was not performed for Subject 003 of treatment group A at any visit and therefore was not analyzed.
  Chest X-ray was performed for Subjects 001, 002, 004, and 005. There was not found to be any improvement of respiratory symptoms across all participants.
  Not enough data to draw statistical inferences between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A | Treatment Group B- HFCC and Cough Assist
Number analyzed (Participants) | 0 | 4
Participants | 0 | 0

2. Primary Outcome: Number of Subjects With Improved Respiratory Symptoms As Shown By Lung Ventilation Scan Between Baseline and End of Study
Description: A nuclear scanning test commonly used to detect abnormalities in air flow. A radioactive tracer gas or mist is inhaled into the lungs. Pictures from the scan indicate areas of the lungs that are not receiving enough air or that retain too much air. Areas of the lung that retain too much air are brighter spots on the film and areas not receiving enough air are dark. Lung scan performed at each study visit. Investigator looked at clinical impression of lung scan to be normal versus abnormal. If there was indication of decreased ventilation, this indicated a worsening of subject's respiratory symptoms. If subject's lung scan impression remained the same and continually normal, this indicated no change in respiratory symptoms.
Time Frame: 1 time at screening/baseline and then at the month 1, month 3, and month 6 study visit for a total of 4 lung ventilation scans over 6 months.
Population: Lung scan was not performed for Subject 003 of treatment group A at any visit and therefore was not analyzed.
  Lung scan was performed for Subjects 001, 002, 004, and 005. There was not found to be any improvement of respiratory symptoms across all participants.
  Not enough data to draw statistical inferences between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A - HFCC Only | Treatment Group B- HFCC and Cough Assist
Number analyzed (Participants) | 0 | 4
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Increased McGill Single Item Quality of Life Scale Question Between Baseline and End of Study
Description: Assess the improvement of/ rate of deterioration of the subject's quality of life from baseline to end of study on a rated scale of 1 to 10.
Time Frame: 1 time at screening/baseline and then at the month 1, month 3, and month 6 study visit for a total of 4 questionnaires over 6 months.
Population: Treatment Group A subject 003 did not complete study. Treatment Group B subjects 001 and 005 were only subjects to complete study and reported upward trend of McGill Quality of Life Scale.
  Not enough data to draw statistical inferences between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A - HFCC Only | Treatment Group B- HFCC and Cough Assist
Number analyzed (Participants) | 0 | 2
Participants | 0 | 2

4. Primary Outcome: Number of Participants With Improved Forced Vital Capacity (FVC) Between Baseline and End of Study
Description: Spirometry will be used to measure FVC. It is the most common of the pulmonary function tests and measures lung function, specifically the measurement of the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled.
Time Frame: 1 time at screening/baseline and then at the month 1, month 3, and month 6 study visit for a total of 4 testing sessions over 6 months.
Population: Treatment Group A subject 003 did not complete study. Treatment Group B subjects 001 and 005 were only subjects to complete study and there was a worsening of FVC values for both subjects.
  Not enough data to draw statistical inferences between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A - HFCC Only | Treatment Group B- HFCC and Cough Assist
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Improved Maximal Inspiratory Pressure (MIP) Between Baseline and End of Study
Description: Spirometry will be used to measure MIP. It is the most common of the pulmonary function tests and measures lung function, specifically the measurement of the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled.
Time Frame: as for outcome 4
Population: Treatment Group A subject 003 did not complete study. Treatment Group B subjects 001 and 005 were only subjects to complete study and there was a worsening of MIP values for both subjects.
  Not enough data to draw statistical inferences between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A - HFCC Only | Treatment Group B- HFCC and Cough Assist
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Improved Diffusion Capacity Between Baseline and End of Study
Description: Spirometry will be used to measure Diffusion Capacity. It is the most common of the pulmonary function tests and measures lung function, specifically the measurement of the amount (volume) and/or speed (flow) of air that can be inhaled and exhaled.
Time Frame: as for outcome 4
Population: Treatment Group A subject 003 did not complete study. Treatment Group B subjects 001 and 005 were only subjects to complete study and there was a worsening of diffusion capacity values for subject 005 and an improvement of subject 005 from 23.1 ml/mmHg/min to 28.7 ml/mmHg/min Not enough data to draw statistical inferences between groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group A - HFCC Only | Treatment Group B- HFCC and Cough Assist
Number analyzed (Participants) | 0 | 2
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 25.7 weeks
Arm/Group | Treatment Group A - HFCC Only | Treatment Group B- HFCC and Cough Assist
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group A - HFCC Only (N=1) | Treatment Group B- HFCC and Cough Assist (N=4)
Death due to respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient with ALS died due to respiratory insufficiency during study

LIMITATIONS AND CAVEATS:
Data too limited to address the aims and perform statistical analyses between the groups. 5 subjects were enrolled, only two completed the study, and the one that was randomized for HFCC only did not have any follow up visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT02682030/Prot_SAP_000.pdf